CLINICAL TRIAL: NCT00293982
Title: The Influence of Expectations on Patient Satisfaction in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CHW 04/22, HRRC 086-04
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2006-02-20 (Estimated); Status verified 2005-02

CONDITIONS: Patient Satisfaction
Keywords: Patient satisfaction; Patient expectations; Pediatric emergency department
MeSH Terms: conditions — Patient Satisfaction

INTERVENTIONS:
Behavioral: Physician knowledge of parental expectations for the visit

SUMMARY:
The purpose of this study is to determine whether physician knowledge of parental pre-visit expectations improves patient satisfaction in the pediatric emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child less than or equal to 18 years of age

Exclusion Criteria:

* Inability to understand the English language surveys

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 948
Dates: Start 2004-06; Study Completion 2005-08

PRIMARY OUTCOMES:
Patient satisfaction as measured by:
1. ratings of overall care
2. willingness to recommend the ED

SECONDARY OUTCOMES:
Ratings of degree to which expectations were met

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Spahr, MD, Principal Investigator — Medical College of Wisconsin; David C Brousseau, MD, MS, Study Director — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States